CLINICAL TRIAL: NCT05331430
Title: Effectiveness of Dry Needling and Stretching on Joint Range and Myofascial Pain at the Cervical Level in People With Fibromyalgia.
Brief Title: Effectiveness of Dry Needling and Stretching in People With Fibromyalgia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Angel Martínez Carrasco, Clinical Professor PhP, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JQR-2022-01
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Dry Needling; Stretch; Fibromyalgia
Keywords: Dry needling; Stretch; Fibromyalgia; Physical Therapy
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Masked participants. Masked data analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1: Dry needling on cervical trigger point (Experimental): Dry needling of the trigger point of the upper fibres of the trapezius muscle. Using the Hong technique.
  Interventions: Other: Dry needling on cervical trigger point
- Experimental group 2: Trapezius muscle stretch (Experimental): Manual passive stretching of the upper trapezius muscle fibres.
  Interventions: Other: Dry needling on cervical trigger point
- Control group: Informative talks (No Intervention): Informative talks on breathing techniques, relaxation techniques and posture hygiene.

INTERVENTIONS:
Other: Dry needling on cervical trigger point — One experimental group will receive dry needling treatment on the upper trapezius fibres using the Hong technique and the other experimental group will receive passive muscle stretching treatment on the upper trapezius fibres.
  Other Names: Trapezius muscle stretch
  Arms: Experimental group 1: Dry needling on cervical trigger point; Experimental group 2: Trapezius muscle stretch

SUMMARY:
Effectiveness of dry needling and stretching on joint range and myofascial pain at the cervical level in people with fibromyalgia

DETAILED DESCRIPTION:
A randomised clinical trial will be conducted in which there will be 3 groups. One control group and 2 experimental groups; one of them will undergo dry needling of the upper trapezius fibres and the other will undergo passive stretching of the upper trapezius fibres. Both groups will have the joint range of cervical lateral tilt, pain measurement by algometer and visual analogue scale (VAS) measured. All these measurements will be taken before and after treatment. The participants of the study will be people who have been diagnosed with fibromyalgia at least 6 months before the start of the study, who are members of the FIBROFAMUR association. Association of Fibromyalgia, Chronic Fatigue, Rheumatic and Musculoskeletal Diseases of Murcia. The data collected will be: socio-demographic data, age, sex, measurement of cervical joint range using a goniometer and measurement of pain using an algometer and visual analogue scale (VAS). As undesirable effects, in exceptional cases, the dry needling technique may produce residual discomfort in the puncture area that may last between 1 and 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of fibromyalgia at least six months before the start of the study.
* Be of legal age.
* Report at least one episode of neck pain in the last six months.

Exclusion Criteria:

* Surgical interventions or scars at cervical level.
* Dizziness or vertigo.
* Dermatological problems.
* Severe psychiatric disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Goniometer measurement | One month
  Measurement of the joint range of the contralateral cervical tilt using a goniometer. Measurement of the lateral tilt range in degrees.Values may vary from zero to 45 degrees.
Measurement of pain with an algometer. | One month
  Measurement of cervical myofascial trigger point pain with an algometer. Measurement of pain in kilograms per square centimetre. Values may vary from zero to 10 kilograms.
Visual analogue scale (VAS) | One month
  Measurement of the degree of pain using the visual analogue scale. Measured from zero to ten, zero corresponds to no pain and ten corresponds to worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Martínez Carrasco, PhD, Study Director — Universidad de Murcia; Jose Quereda Ruiz, Graduated, Principal Investigator — Universidad de Murcia
Locations (1):
- Universidad de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No